CLINICAL TRIAL: NCT06148233
Title: CSF1R PET Probe [18F]CSF-23 in Alzheimer's Disease Brain Imaging
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, YiHui Guan, Professor, Huashan Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KY2023-780
Record Dates: First submitted 2023-11-19; First posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Positron Emission Tomography; Alzheimer Disease; Neurodegenerative Diseases
MeSH Terms: conditions — Alzheimer Disease; Neurodegenerative Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with Alzheimer's Disease (Experimental): AD subjects recruited from geriatric wards or memory clinics.
  Interventions: Radiation: [18F]CSF-23
- Cognitively normal control group (Experimental): Cognitively normal subjects recruited from the community
  Interventions: Radiation: [18F]CSF-23

INTERVENTIONS:
Radiation: [18F]CSF-23 — Intravenous injection of 1.8 MBq [0.05MCi]/kg of [18F]CSF-23 in a single dose.

SUMMARY:
To explore the diagnostic value of [18F]CSF-23 brain imaging for CSF1R expression in Alzheimer's disease. PET imaging with this PET tracer was used to assess the role and expression of CSF1R in AD and to evaluate the level and safety of abnormal present imaging.

ELIGIBILITY:
Inclusion Criteria:

* Non-diseased controls:

  1. Between 60 and 80 years of age; gender is not limited.
  2. Cognitively normal as determined by the investigator through testing, with an MMSE score greater than 25 and no cognitive domain impairment. They had a negative Aβ image.
  3. No neurological diseases, major chronic diseases, malignant tumors, or acute infectious diseases, as determined by the investigator.
  4. Written informed consent must be signed by the subject or his/her legal guardian or caregiver.
  5. Blood routine: white blood cell count (WBC) 4~10×109/L; platelet (PLT) 100~300×109/L; hemoglobin (HB) 120~160 g/L; renal function: serum creatinine less than or equal to the upper limit of the normal range; hepatic function: bilirubin, AST (SGOT)/ALT (SGPT) less than or equal to the upper limit of the normal range; Electrocardiogram: no significant abnormalities.
  6. No neurological diseases, major chronic diseases, malignant tumors, or acute infectious diseases, as confirmed by the investigator; no family history of neurodegenerative movement disorders, and no family history of neurological disorders related to movement disorders.
  7. Willingness and ability to cooperate with all programs of this study.

AD patients:

1. Age between 60 and 80 years old; gender is not limited.
2. Patients meet the 2011 NIA-AA diagnostic criteria for red AD patients and have positive Aβ images.
3. Brain MRI supported the diagnosis of AD and there was no evidence of other neurological diseases.
4. No neurological diseases, major chronic diseases, malignant tumors or acute infectious diseases, etc., as confirmed by the investigator.
5. Written informed consent must be signed by the subject or his/her legal guardian or caregiver.
6. Blood routine: white blood cell count (WBC) 4~10×109/L; platelet (PLT) 100~300×109/L; hemoglobin (HB) 120~160 g/L; renal function: serum creatinine less than or equal to the upper limit of the normal range; hepatic function: bilirubin, AST (SGOT)/ALT (SGPT) less than or equal to the upper limit of the normal range; ECG: no significant abnormalities.
7. No neurological diseases, major chronic diseases, malignant tumors, or acute infectious diseases, as confirmed by the investigator; no family history of neurodegenerative movement disorders, and no family history of neurological disorders related to movement disorders.
8. Willingness and ability to cooperate with all programs of this study.

Exclusion Criteria:

* Subjects meeting any of the following criteria will be excluded from the study:

  1. Severe hepatic or renal insufficiency;
  2. Participation in other research protocols or clinical care within the past year, in addition to the radiation exposure expected from participation in this clinical study, which has resulted in radiation exposure in excess of an effective dose of 50 mSv.
  3. Liver function: bilirubin, AST(SGOT)/ALT(SGPT) less than or equal to the upper limit of the normal range.
  4. History of serious surgery in the last month.
  5. Participation in other clinical trials during the same period.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-06-16 (Estimated); Study Completion 2024-09-14 (Estimated)

PRIMARY OUTCOMES:
Complete PET imaging | 90mins from time of injection
  To assess the diagnostic value of [18F]CSF-23 brain imaging for CSF1R expression in Alzheimer's disease.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Xie, PhD, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital, Shanghai, China